CLINICAL TRIAL: NCT04833309
Title: Effectiveness and Safety of Pharmacopunture Therapy for Chronic Low Back Pain: A Pragmatic Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director of Jaseng Spine and Joint Research Institute, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-02
Record Dates: First submitted 2021-04-04; First posted 2021-04-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacopuncture therapy (Experimental): Pharmacopuncture will be administered to the subjects in the pharmacopuncture therapy group. The physicians will choose the specific type and volume of pharmacopuncture according to participants' conditions.
  Interventions: Procedure: pharmacopuncture therapy
- Physical therapy (Active Comparator): Physical therapy will be applied to the subjects in the physical therapy group. The physicians will choose the specific type and volume of pharmacopuncture according to participants' conditions.
  Interventions: Procedure: physical therapy

INTERVENTIONS:
Procedure: pharmacopuncture therapy — The procedure will be implemented to participants twice a week for total 5 weeks. The specific prescription including type and dosage will be determined according to the physician's choice, and information will be recorded in the case report form retrospectively.
  Arms: Pharmacopuncture therapy
Procedure: physical therapy — The procedure will be implemented to participants twice a week for total 5 weeks. The specific prescription including type and body part will be determined according to the physician's choice, and information will be recorded in the case report form retrospectively.
  Arms: Physical therapy

SUMMARY:
This is a multi-center, 2-arm parallel pragmatic randomized controlled trial that will compare pharmacopuncture therapy with physical therapy for chronic low back pain.

DETAILED DESCRIPTION:
This is a multi-center, 2-arm parallel pragmatic randomized controlled trial that will compare pharmacopuncture therapy with physical therapy for chronic low back pain. Participants who voluntarily signed informed consent form and eligible for the study were randomly assigned in a 1:1 ratio (50:50) for pharmacopuncture therapy group and physical therapy group. Participants of each group will receive total 5 weeks of intervention. This is a pragmatic randomized controlled trial, so physicians will have medical decision making according to each participant's conditions and choose the specific type and volume of pharmacopuncture and physical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. low back pain for more than 6 months
2. Numeric rating scale (NRS) score for low back pain 5 or more
3. 19-70 years old
4. participants who agreed and signed informed consent form

Exclusion Criteria:

1. Spine metastasis of cancer, acute fracture of spine, or spine dislocation
2. Progressive neurologic deficits or severe neurologic deficits
3. Soft tissue diseases that can induce low back pain (ie. cancer, fibromyalgia, rheumatoid arthritis, gout, etc)
4. Presence of chronic underlying disease which can interfere the efficacy or interpretation (ie. stroke, myocardial infarct, kidney disease, dementia, diabetic neuropathy, epilepsy, etc)
5. Concurrent use of steroids, immunosuppressants, or psychotropic medications
6. Hemorrhagic disease, severe diabetes or taking anticoagulant drug
7. Participants who took NSAIDs or pharmacopuncture within 1 week
8. Pregnant or lactating women
9. Participants who had undergone lumbar surgery within 3 months
10. Participants who had participated in other clinical trial within 1 month, or have plan for participation in other trial during follow up period of this trial
11. Participants who can not write informed consent
12. Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) of low-back pain | week 6
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of low-back pain | week 1, 2, 3, 4, 5, 6, 13, 25
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Numeric rating scale (NRS) of radiating pain in lower extremities | week 1, 2, 3, 4, 5, 6, 13, 25
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Visual analogue scale (VAS) of leg radiating pain | week 1, 2, 3, 4, 5, 6, 13, 25
  Visual analogue scale of radiating leg pain, minimum 0 to maximum 100, which is a higher score means a worse outcome.
Visual analogue scale (VAS) of low-back pain | week 1, 2, 3, 4, 5, 6, 13, 25
  Visual analogue scale of radiating leg pain, minimum 0 to maximum 100, which is a higher score means a worse outcome.
Oswestry Disability Index (ODI) | week 1, 6, 13, 25
  ODI is a functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range is 0 (better outcome) to 100 (worse outcome).
Korean version of the Roland-Morris Disability Questionnaire (RMDQ) | week 1, 6, 13, 25
  The Roland Morris Disability Questionnaire consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). There is no weighting applied to the statements, therefore the score can range from 0 (no disability) to 24 (maximal disability).
Patient Global Impression of Change (PGIC) | week 6, 13, 25
  Participants rate the improvement after treatment on a 7-point Likert scale (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.)
Short Form-12 Health Survey version 2 (SF-12 v2) | week 1, 6, 13, 25
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
EuroQol-5 Dimension (EQ-5D-5L) | week 1, 6, 13, 25
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about)

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD,Ph.D, Study Director — Jaseng Medical Foundation
Locations (4):
- South Korea (4):
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YS, Kim SJ, Park KS, Lee YJ, Yang C, Han CH, Ha IH. A cost-utility analysis of pharmacopuncture versus physiotherapy for chronic low back pain: A multicenter, pragmatic randomized controlled trial. Integr Med Res. 2025 Dec;14(4):101210. doi: 10.1016/j.imr.2025.101210. Epub 2025 Aug 5. PMID 41497196
- [Derived] Park KS, Kim S, Seo JY, Cho H, Lee JY, Lee YJ, Lee J, Kim MJ, Choi YE, Yang CS, Han CH, Ha IH. Effectiveness and Safety of Pharmacopuncture Therapy for Chronic Low Back Pain: A Protocol for a Pragmatic Randomized Controlled Trial. J Pain Res. 2022 Sep 1;15:2629-2639. doi: 10.2147/JPR.S375231. eCollection 2022. PMID 36072909

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04833309/Prot_SAP_000.pdf